CLINICAL TRIAL: NCT07400744
Title: Phase I Study to Compare the Pharmacokinetic Characteristics, Safety, and Immunogenicity (Randomized, Double-blind, Single Dose, Parallel Controlled) of QL2109 With Daratumumab Injection in Healthy Chinese Male Subjects
Brief Title: A Study to Compare the PK , Safety, and Immunogenicity of QL2109 With Daratumumab in Male Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL2109-102
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL2109 (Experimental)
  Interventions: Drug: QL2109
- Darzalex (Active Comparator)
  Interventions: Drug: Darzalex

INTERVENTIONS:
Drug: QL2109 — Recombinant anti-CD38 fully human monoclonal antibody.
  Arms: QL2109
Drug: Darzalex — Daratumumab injection
  Arms: Darzalex

SUMMARY:
The goal of this clinical study is to establish the comparability of the pharmacokinetics and similarity of the safety and immunogenicity profiles of QL2109 and Darzalex following a single intravenous infusion in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. The subject should be a voluntary participant who has understood and signed the ICF.
2. Age ≥ 18 years and ≤ 50 years, male (including the boundary values).
3. Body weight ≥ 55 kilograms (kg), body mass index (BMI) = weight (kg) / height² (m²), with BMI within the range of 18-28 (including the boundary values).
4. The subject agrees to use reliable contraceptive measures (such as abstinence, sterilization surgery, oral contraceptives, injectable contraceptives like medroxyprogesterone, or subcutaneous contraceptive implants) for themselves and their partner during the study and for 6 months after the trial drug infusion.
5. No history of diseases, or any past medical history abnormalities are deemed clinically insignificant and judged by the study physician to have no impact on the trial.

Exclusion Criteria:

1. Individuals with a history or current diagnosis of any clinically significant disease that may interfere with the trial results, including but not limited to disorders of the circulatory, endocrine, nervous, digestive, respiratory, hematological, immunological, psychiatric, or metabolic systems, or those with clinically significant allergic reactions or allergic predisposition, angioedema, interstitial pneumonia, or acute respiratory distress syndrome.
2. Individuals with acute, chronic, or potential infectious diseases within 1 month prior to dosing.
3. Individuals with known immune system disorders (autoimmune diseases or immunodeficiency diseases), including but not limited to autoimmune hemolytic anemia.
4. Individuals with ocular diseases, including a history of intraocular surgery or laser eye surgery.
5. Individuals with a history of localized cutaneous herpes zoster within 6 months prior to dosing.
6. Individuals with disseminated cutaneous herpes zoster or herpes zoster involving the central nervous system, either currently or historically.
7. Individuals with a positive blood group antibody screening (indirect antiglobulin test).
8. Individuals who have used monoclonal antibodies, cell therapies, or similar treatments within 6 months prior to dosing, or have previously received daratumumab or its analogues, or drugs targeting CD38.
9. Individuals who have taken any medications (except premedication for QL2109 injection/DARZALEX®) within 2 weeks prior to dosing, including prescription drugs, over-the-counter drugs, and herbal medicines.
10. Individuals with a history of drug or food allergies, including allergies to any drug or excipient used in the clinical trial.
11. Individuals with a history of needle or blood phobia, or difficulty with venous blood collection (e.g., history of difficult blood draws or symptoms/signs indicating intolerance to venipuncture).
12. Individuals who have donated blood or experienced blood loss totaling 200 mL or more within 3 months prior to dosing.
13. Individuals who have participated in any other drug or medical device clinical trials within 3 months prior to dosing (or within 5 half-lives of the investigational drug if the half-life exceeds 3 months).
14. Individuals who have undergone major surgery within 3 months prior to signing the informed consent form (ICF).
15. Individuals who are positive for hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg), and/or hepatitis B core antibody (HBcAb); positive for hepatitis C virus antibody (HCV); positive for Treponema pallidum antibody; or positive for human immunodeficiency virus (HIV) antibody.
16. Individuals with a history of drug abuse or substance dependence, or those with a positive urine drug screen.
17. Individuals who have received live attenuated or live virus vaccines (e.g., Bacille Calmette-Guérin [BCG]) or viral vector vaccines within 12 months prior to the first dose, or plan to receive such vaccines within 12 months after dosing.
18. Individuals who have received other vaccines, such as inactivated vaccines or recombinant subunit vaccines, within 1 month prior to the first dose, excluding the aforementioned live attenuated or live virus vaccines and viral vector vaccines.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
AUC0-∞ | Up to Day 71
  Area under the serum concentration-time curve from time 0 to infinity